CLINICAL TRIAL: NCT04656210
Title: Links Between Diabetes and Cognitive Impairment in Myotonic Dystrophy Type 1 : a Non-conventional MRI Study
Brief Title: Myotonic Dystrophy - Vascular and Cognition
Acronym: DM-VASCOG
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018_31; 2019-A00086-51 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2020-11-23; First posted 2020-12-07 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Myotonic Dystrophy 1; Diabetes; Carbohydrate Intolerance
Keywords: Cerebral atrophy; MRI; cognition; metabolic syndrome; tauopathy
MeSH Terms: conditions — Myotonic Dystrophy; Diabetes Mellitus; Glucose-Galactose Malabsorption; Metabolic Syndrome; Tauopathies | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: MD type 1 normal: patients with type 1 myotonic dystrophy with normal carbohydrate tolerance
  Interventions: Radiation: MRI; Other: neuropsychological tests
- Group 2: MD type 1 Diabetes: patients with type 1 myotonic dystrophy with diabetes. Patients with carbohydrate intolerance ("pre-diabetes") who became diabetic at 3 years of age will be divided into Group 2.
  Interventions: Radiation: MRI; Other: neuropsychological tests

INTERVENTIONS:
Radiation: MRI — Non conventional MRI (35 minutes)
Other: neuropsychological tests — Standardized and quantified neuropsychological assessment

SUMMARY:
The cognitive disorders of adult forms of myotonic dystrophies type 1 are heterogeneous (impairment of executive functions, visio construction and theory of the mind, which can progress to the stage of dementia). Nevertheless, patients have very different degrees of cognitive impairment. Expansion of CTG triplets disrupts the alternative splicing of mRNAs of various proteins, including the insulin receptor and Tau protein. Type 2 diabetes, associated with peripheral insulin resistance, is therefore common in this pathology.

Type 2 diabetes,could to explain the cognitive impairment of patients, through the accelerated development of brain lesions (especially tauopathy and cerebral atrophy).

ELIGIBILITY:
Inclusion Criteria:

* Molecularly proven type 1 myotonic dystrophy
* Voluntary, having given informed consent
* Socially insured patient
* Patient willing to comply with all study procedures and duration (3 hours + MRI 35 minutes)
* Patient insured under the French social security system
* Signed consent form

Exclusion Criteria:

* Neurological history other than neuropathy: epilepsy, stroke, dementia
* Pregnancy or breastfeeding or woman of childbearing age without effective contraception (a pregnancy test will be done)
* Contra indication to MRI
* Person under guardianship or curators
* Persons of full age deprived of their liberties by a judicial or administrative decision
* Major comorbidity considered as a contraindication by the investigator (cancer, unstable angina, etc.).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with DM type 1 monitored annually by the Neuromuscular Disease Reference Centre
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2024-10-13 (Actual); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Atrophy difference based on two cerebral MRI volumetries | at 4 years
  difference between initial MRI and 4-year MRI

SECONDARY OUTCOMES:
changes in scores at 4-year neuropsychological assessment of inclusion | At baseline at 4 years
  difference between initial assessment and 4-year assessment
changes in tau biomarkers in blood at 4 years of inclusion | At baseline at 4 years
  difference between initial and 4-year dosing
changes in amyloid biomarkers in blood at 4 years of inclusion | At baseline at 4 years
  difference between initial and 4-year dosing

CONTACTS AND LOCATIONS:
Overall Officials: Céline TARD, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hopital Roger Salengro, CHU Lille, Lille, France